CLINICAL TRIAL: NCT02242409
Title: A Phase II Study of Gemcitabine and Nanoparticle-Bound Paclitaxel as Second Line Therapy in Patients With Metastatic Pancreatic Cancer
Brief Title: Study of Gemcitabine and Abraxane for Pancreas Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Testing of combination no longer relevant
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 2013-0138
Record Dates: First submitted 2014-09-12; First posted 2014-09-17 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Pancreatic Cancer
Keywords: Metastatic pancreatic cancer; Second Line treatment; Gemcitabine; Nab-paclitaxel
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine/abraxane (Experimental): Gemcitabine and Abraxane
  Interventions: Drug: Gemcitabine and Abraxane

INTERVENTIONS:
Drug: Gemcitabine and Abraxane — Gemcitabine 1000 mg/m2 followed by abraxane 125 mg/m2 administered intravenously on days 1, 8, and 15 every 28 days
  Other Names: Gemzar; nanoparticle-bound paclitaxel; Nab-paclitaxel

SUMMARY:
A Phase II trial of gemcitabine plus nab-paclitaxel in the second line setting

DETAILED DESCRIPTION:
This is an open label Phase II study to evaluate the clinical activity of the combination of gemcitabine and nab-paclitaxel (abraxane) as second line treatment in patients with metastatic pancreatic cancer who have received non-gemcitabine-based chemotherapy in the first line setting. All patients will receive both drugs on Days 1, 8, 15 every 28 days. The hypothesis is that this combination will have a 4-month progression free survival of 70% or higher.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic adenocarcinoma of the pancreas
* Progression on first line non-gemcitabine based therapy for metastatic or relapsed disease
* Radiographically measurable or evaluable disease
* Age >/= 18 years
* ECOG performance status 0-2
* Adequate hepatic, bone marrow and renal function

Exclusion Criteria:

* Prior gemcitabine-based chemotherapy in the first line setting
* No active severe infection, or known chronic infection with HIV or hepatitis B virus
* No cardiovascular disease problems including unstable angina, therapy for life-threatening ventricular arrhythmia, or myocardial infarction, stroke, or congestive heart failure within the last 6 months
* No women who are pregnant or breastfeeding, and no women of childbearing potential without using dual forms of contraception
* Patients with known CNS metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to gemcitabine or nab-paclitaxel
* Anticipated patient survival under 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
4 month progression free survival | 2.5 years
  The proportion of patients at 4 months from study entry with progression or death

SECONDARY OUTCOMES:
Disease control rate | 2.5 years
  Confirmed classification of stable disease, partial response or complete response by RECIST 1.1 criteria
Progression Free Survival | 2.5 years
  The time in days from study entry until progression or death
Overall Survival | 3 years
  The time in days from study entry until death

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pishvaian, MD PhD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia, United States